CLINICAL TRIAL: NCT01767896
Title: Phase III Study of ASP7374 -Approved Egg-derived Vaccine Controlled, Double-blind, Parallel Group Study in Elderly Subjects
Brief Title: Phase-3 Study of ASP7374, Cell-culture-derived Influenza Vaccine
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: UMN Pharma Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: 7374-CL-0103
Record Dates: First submitted 2013-01-11; First posted 2013-01-15 (Estimated); Last update posted 2017-09-29 (Actual); Status verified 2017-09

CONDITIONS: Influenza
Keywords: Influenza vaccine
MeSH Terms: conditions — Influenza, Human

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- ASP7374 group (Experimental): cell-culture-derived vaccine group
  Interventions: Biological: ASP7374
- TIV group (Active Comparator): approved egg-derived TIV group
  Interventions: Biological: approved egg-derived TIV

INTERVENTIONS:
Biological: ASP7374 — subcutaneous (sc)
  Arms: ASP7374 group
Biological: approved egg-derived TIV — subcutaneous (sc)
  Other Names: Influenza HA vaccine "SEIKEN"
  Arms: TIV group

SUMMARY:
The purpose of this study is to compare immunogenicity and safety of ASP7374 (cell-culture derived influenza vaccine) with those of approved egg-derived trivalent inactivated vaccine (TIV) in elderly subjects.

ELIGIBILITY:
Inclusion Criteria:

* Medically stable, as judged on the basis of history and concurrent diseases
* Subject understands procedure of the protocol and is willing to comply with the protocol

Exclusion Criteria:

* Scheduled to receive another vaccine during the study
* Received influenza HA vaccine within 180 days prior to screening
* Received or scheduled to receive a live vaccine within 28 days prior to vaccination with the study vaccine, and received or scheduled to receive an inactivated vaccine or a toxoid within 7 days prior to vaccination with the study vaccine
* Diagnosis of immune deficit in the past, has a family member (within the third degree of kinship) with a diagnosis of congenital immunodeficiency syndrome
* Received one of the following medications or treatment prior to vaccination with the study vaccine: Interferon formulation, drugs which affect the immune system, corticosteroids, G-CSF, M-CSF, human immunoglobulin products, blood products
* History of anaphylactic shock or an allergic reaction such as generalized eruption due to food or drug (including vaccines) allergies, fever ≥39.0°C within 2 days after the previous vaccination (influenza vaccine and others)
* History of seizures
* History of Guillain-Barre syndrome or acute disseminated encephalomyelitis (ADEM)
* Confirmed diagnosis of influenza within 84 days prior to screening test
* Body temperature of ≥37.5°C on Day 1 (before vaccination)
* Immunological tests reveal positive HBs antigen, HCV antibody, and HIV antigen and/or antibody

Min Age: 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Older Adult
Enrollment: 1020 (Actual)
Dates: Start 2012-10; Primary Completion 2013-03 (Actual); Study Completion 2013-03 (Actual)

PRIMARY OUTCOMES:
seroconversion rate of hemoagglutination inhibition (HI) antibody titer | Day 29
  evaluated for A/H1N1, A/H3N2, and B
geometric mean titer (GMT) of HI antibody titer | Day 29
  evaluated for A/H1N1, A/H3N2, and B

SECONDARY OUTCOMES:
seroprotection rate of HI antibody titer | Day 29
  evaluated for A/H1N1, A/H3N2, and B
GMT ratio of HI antibody titer | Day 1 and Day 29
  evaluated for A/H1N1, A/H3N2, and B
seroconversion rate of neutralizing antibody titer | Day 29
  evaluated for A/H1N1, A/H3N2, and B
seroprotection rate of neutralizing antibody titer | Day 29
  evaluated for A/H1N1, A/H3N2, and B
GMT of neutralizing antibody | Day 29
  evaluated for A/H1N1, A/H3N2, and B
GMT ratio of neutralizing antibody | Day 1 and Day 29
  evaluated for A/H1N1, A/H3N2, and B

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Astellas Pharma Inc
Locations (3):
- Japan (3):
  - Kansai
  - Kantou
  - Kyushu